CLINICAL TRIAL: NCT00276952
Title: Phase 2 Study of Treatment of Chronic Tension-Type Headache Using Gonyautoxins
Brief Title: Gonyautoxin in the Treatment of Chronic Tension-Type Headache
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chile (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HCUCH-NL-GTX-002
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2006-01-13 (Estimated); Status verified 2005-09

CONDITIONS: Tension-Type Headache
Keywords: Gonyautoxins; Tension-type Headache; Human Treatment
MeSH Terms: conditions — Tension-Type Headache | interventions — gonyautoxins

INTERVENTIONS:
Drug: Gonyautoxin

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of Gonyautoxin 2/3 epimers in the treatment of patients diagnosed with chronic tensional-type headache in accordance with International Headache Society guidelines

DETAILED DESCRIPTION:
Gonyautoxin are phycotoxins, whose molecular mechanism of action is a reversible block of the voltage-gated sodium channels at neuronal level. They are axonal conduction blockers impeding nerve impulse propagation. In order to evaluate the clinical efficacy of Gonyautoxin 2/3 epimers in the treatment of patients diagnosed with chronic tensional-type headache, the patients were locally injected with placebo versus Gonyautoxin following a painful spots injection standarized protocol

ELIGIBILITY:
Inclusion Criteria:

* Chronic tensional-type headache patients according to the International Headache Society criteria: patients with headache of a pressing or tightening quality with episodic frequency above 15 days a month
* Refractory to conventional treatments such as, orally administered analgesics, systemic muscular relaxant, corticoids and antidepressant like Amytriptiline
* Treated and controlled in the University Hospital Neurology Clinic over 2 years with duration of symptoms over 3 years

Exclusion Criteria:

* Pregnancy
* Use of headache prophylactic treatment a month prior to infiltration
* Myasthenic syndromes
* Muscular dystrophies
* Inflammatory myopathies
* Acute and chronic polineuropathies
* Use of psychotropic substances 24-hour before infiltration
* Anticoagulant treatment
* terminal illnesses (AIDS, cancer)
* drugs or alcohol abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27
Dates: Start 2004-09; Study Completion 2005-08

PRIMARY OUTCOMES:
a) Drop off in the patient acute headache pain (2 minutes, weekly for 20 weeks)
b) Number of days without headache pain following infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Lagos, PhD, Principal Investigator — Faculty of Medicine University of Chile
Locations (1):
- Departament of Neurology and Neurosurgery, Hospital Clínico Universidad de Chile., Santiago, Santiago Metropolitan, Chile